CLINICAL TRIAL: NCT03905317
Title: A Single-Armed Phase II Study of Radiation and Bevacizumab Maintenance Therapy for Oligometastasis of Lung Adenocarcinoma With Negative Driver Gene
Brief Title: Bevacizumab and Radiotherapy for Oligometastasis of Lung Adenocarcinoma With Negative Driver Gene
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1047
Record Dates: First submitted 2019-03-15; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-02

CONDITIONS: Lung Adenocarcinoma
Keywords: bevacizumab; chemoradiotherapy; Oligometastasis of lung adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab (Experimental): The patients receive SBRT radiotherapy for the primary (if any) and metastatic lesions or divided radiotherapy with or without concurrent chemotherapy.Bevacizumab maintenance therapy starts 1-2 months later after the chemotherapy.The recommended dose for intravenous infusion is 15mg/kg body weight, and the drug is given every 3 weeks until disease progression or intolerable toxicity occurs.
  Interventions: Drug: Bevacizumab Injection; Radiation: chest radiation; Drug: concurrent chemotherapy

INTERVENTIONS:
Drug: Bevacizumab Injection — Bevacizumab maintenance therapy starts 1-2 months later after the chemotherapy.The recommended dose for intravenous infusion is 15mg/kg body weight, and the drug is given every 3 weeks until disease progression or intolerable toxicity occurs.
Radiation: chest radiation — The patients receive SBRT radiotherapy for the primary (if any) and metastatic lesions or divided radiotherapy with or without concurrent chemotherapy.
Drug: concurrent chemotherapy — weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡) concurrent with chest radiation

SUMMARY:
This prospective phase II study is determined to explore the efficacy and safety of radiotherapy and bevacizumab maintenance therapy for oligometastatic lung adenocarcinoma with negative driver genes

DETAILED DESCRIPTION:
This prospective phase II study is determined to explore the efficacy and safety of radiotherapy and bevacizumab maintenance therapy for oligometastatic lung adenocarcinoma with negative driver genes.

The patients receive SBRT radiotherapy for the primary (if any) and metastatic lesions or divided radiotherapy with or without concurrent chemotherapy.Bevacizumab maintenance therapy starts 1-2 months later after the chemotherapy.The recommended dose for intravenous infusion is 15mg/kg body weight, and the drug is given every 3 weeks until disease progression or intolerable toxicity occurs. Toxicities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of lung adenocarcinoma with negative driver gene including EGFR and ALK.
* Simultaneous oligometastasis, or oligometastasis which occurs after treatment of stage i-iii lung adenocarcinoma (1-5 metastases)
* Oligometasis confirmed by CT, brain MR, bone ECT or PETCT within 30 days before enrollment.

Exclusion Criteria:

* ≥18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Organ and bone marrow functions are normal within the first 30 days of enrollment, including: • AST, ALT≤ 2.5*ULN or ≤5*ULN (with liver metastasis); • TBil ≤ 1.5 ULN • neutrophils absolute value ≥500 cells/mm3 • creatinine clearance ≥45 mL/min ;• platelets≥50,000 cells/mm3.
* Negative pregnancy test 1 week before enrollment for women of childbearing age.
* Patients with concurrent oligostasis should have received at least 4 courses of first-line chemotherapy, and SD or PR should be evaluated after chemotherapy;
* Patients with stage i-iii lung adenocarcinoma with oligo-metastasis after treatment who have previously received systemic chemotherapy (such as concurrent radiotherapy chemotherapy or postoperative adjuvant chemotherapy) are admitted to the group;
* Patients who have received brain radiation therapy due to brain metastasis are admitted to the group.
* The baseline is the exsiting of measurable lesions, and the metastatic lesions are treated with local radiotherapy;The number of metastases defines as:
* - A) two metastatic lesions are identified when bilateral adrenal glands have lesions;
* - B) two consecutive vertebral lesions and paravertebral lesions within 6cm can be considered as one metastatic lesion, and the lesions of non-continuous vertebral body should be counted separately;
* - C) the adjacent lesions in the liver, lung and mediastinum can be considered as a metastatic lesion if one isocentric irradiation can be used;
* For simultaneous oligostasis, the feasibility of primary focus radiotherapy should be evaluated, and the primary focus must be capable of receiving radiotherapy before being enrolled;For the primary lesion, SBRT or fractionated radiotherapy can be applied according to the site and surrounding invasion.
* For the heterogeneous oligometastasis of the primary lesion that has received surgery or local radiotherapy, the feasibility of local radiotherapy should be evaluated when the local recurrence lesion occurs, and the local recurrence lesion can be treated with subdivided radiotherapy or SBRT before inclusion;
* Patients with intracranial metastasis are allowed to be enrolled, but the intracranial lesions should be treated in advance and be in a stable state, and the number of intracranial lesions should be counted within the number of metastases.
* Patients should be enrolled within 35 days after the last systemic treatment;
* Patients and their family signed the informed consents.

Exclusion Criteria:

* Lung squamous carcinoma.
* The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava).
* The tumor is associated with a cavity over 2cm in diameter.
* Bleeding tendency or coagulation disorder.
* Patients with hemoptysis (1/2 teaspoon blood/day) within 1 month.
* Full-dose anticoagulation therapy was used within the past 1 month.
* Severe vascular disease occurred within 6 months.
* Gastrointestinal fistula, perforation or abdominal abscess occurred within 6 months.
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months.
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg).
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours.
* Urine protein 3-4+, or 24h urine protein quantitative >1g.
* ≥Degree 3 esophagitis after chemoradiotherapy has not recovered.
* The investigator does not consider the participant to be eligible for this study.
* Metastatic lesions involving esophagus, stomach, small intestine or mesenteric lymph nodes;
* The metastatic lesion is adjacent to the primary radiation range, and the radiotherapy physician cannot tolerate the secondary radiotherapy;
* Malignant pleural effusion without obvious remission after first-line chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
PFS | 3-year
  Progression-free survival in patients

SECONDARY OUTCOMES:
OS | 3-year
  overall survival in patients
response rate | 3-year
rate of grade 3-4 radiation esophagitis | 3-year
rate of grade 3-4 radiation pneumonitis | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Albain KS, Crowley JJ, LeBlanc M, Livingston RB. Survival determinants in extensive-stage non-small-cell lung cancer: the Southwest Oncology Group experience. J Clin Oncol. 1991 Sep;9(9):1618-26. doi: 10.1200/JCO.1991.9.9.1618. PMID 1651993
- [Background] Parikh RB, Cronin AM, Kozono DE, Oxnard GR, Mak RH, Jackman DM, Lo PC, Baldini EH, Johnson BE, Chen AB. Definitive primary therapy in patients presenting with oligometastatic non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):880-7. doi: 10.1016/j.ijrobp.2014.04.007. Epub 2014 May 24. PMID 24867533
- [Background] Lewis SL, Porceddu S, Nakamura N, Palma DA, Lo SS, Hoskin P, Moghanaki D, Chmura SJ, Salama JK. Definitive Stereotactic Body Radiotherapy (SBRT) for Extracranial Oligometastases: An International Survey of >1000 Radiation Oncologists. Am J Clin Oncol. 2017 Aug;40(4):418-422. doi: 10.1097/COC.0000000000000169. PMID 25647831
- [Background] Xanthopoulos EP, Handorf E, Simone CB 2nd, Grover S, Fernandes AT, Sharma S, Corradetti MN, Evans TL, Langer CJ, Mitra N, Shah A, Apisarnthanarax S, Lin LL, Rengan R. Definitive dose thoracic radiation therapy in oligometastatic non-small cell lung cancer: A hypothesis-generating study. Pract Radiat Oncol. 2015 Jul-Aug;5(4):e355-63. doi: 10.1016/j.prro.2014.11.006. Epub 2015 Jan 31. PMID 25649540
- [Background] Iyengar P, Kavanagh BD, Wardak Z, Smith I, Ahn C, Gerber DE, Dowell J, Hughes R, Abdulrahman R, Camidge DR, Gaspar LE, Doebele RC, Bunn PA, Choy H, Timmerman R. Phase II trial of stereotactic body radiation therapy combined with erlotinib for patients with limited but progressive metastatic non-small-cell lung cancer. J Clin Oncol. 2014 Dec 1;32(34):3824-30. doi: 10.1200/JCO.2014.56.7412. Epub 2014 Oct 27. PMID 25349291
- [Background] Collen C, Christian N, Schallier D, Meysman M, Duchateau M, Storme G, De Ridder M. Phase II study of stereotactic body radiotherapy to primary tumor and metastatic locations in oligometastatic nonsmall-cell lung cancer patients. Ann Oncol. 2014 Oct;25(10):1954-1959. doi: 10.1093/annonc/mdu370. Epub 2014 Aug 11. PMID 25114022
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Brodowicz T, Krzakowski M, Zwitter M, Tzekova V, Ramlau R, Ghilezan N, Ciuleanu T, Cucevic B, Gyurkovits K, Ulsperger E, Jassem J, Grgic M, Saip P, Szilasi M, Wiltschke C, Wagnerova M, Oskina N, Soldatenkova V, Zielinski C, Wenczl M; Central European Cooperative Oncology Group CECOG. Cisplatin and gemcitabine first-line chemotherapy followed by maintenance gemcitabine or best supportive care in advanced non-small cell lung cancer: a phase III trial. Lung Cancer. 2006 May;52(2):155-63. doi: 10.1016/j.lungcan.2006.01.006. Epub 2006 Mar 29. PMID 16569462
- [Background] Gerber DE. Maintenance therapy for advanced lung cancer: who, what, and when? J Clin Oncol. 2013 Aug 20;31(24):2983-90. doi: 10.1200/JCO.2012.48.5201. Epub 2013 Jul 8. PMID 23835703
- [Background] Ciuleanu T, Brodowicz T, Zielinski C, Kim JH, Krzakowski M, Laack E, Wu YL, Bover I, Begbie S, Tzekova V, Cucevic B, Pereira JR, Yang SH, Madhavan J, Sugarman KP, Peterson P, John WJ, Krejcy K, Belani CP. Maintenance pemetrexed plus best supportive care versus placebo plus best supportive care for non-small-cell lung cancer: a randomised, double-blind, phase 3 study. Lancet. 2009 Oct 24;374(9699):1432-40. doi: 10.1016/S0140-6736(09)61497-5. Epub 2009 Sep 18. PMID 19767093
- [Background] Paz-Ares L, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. Maintenance therapy with pemetrexed plus best supportive care versus placebo plus best supportive care after induction therapy with pemetrexed plus cisplatin for advanced non-squamous non-small-cell lung cancer (PARAMOUNT): a double-blind, phase 3, randomised controlled trial. Lancet Oncol. 2012 Mar;13(3):247-55. doi: 10.1016/S1470-2045(12)70063-3. Epub 2012 Feb 16. PMID 22341744
- [Background] Fidias PM, Dakhil SR, Lyss AP, Loesch DM, Waterhouse DM, Bromund JL, Chen R, Hristova-Kazmierski M, Treat J, Obasaju CK, Marciniak M, Gill J, Schiller JH. Phase III study of immediate compared with delayed docetaxel after front-line therapy with gemcitabine plus carboplatin in advanced non-small-cell lung cancer. J Clin Oncol. 2009 Feb 1;27(4):591-8. doi: 10.1200/JCO.2008.17.1405. Epub 2008 Dec 15. PMID 19075278
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Reck M, von Pawel J, Zatloukal P, Ramlau R, Gorbounova V, Hirsh V, Leighl N, Mezger J, Archer V, Moore N, Manegold C. Phase III trial of cisplatin plus gemcitabine with either placebo or bevacizumab as first-line therapy for nonsquamous non-small-cell lung cancer: AVAil. J Clin Oncol. 2009 Mar 10;27(8):1227-34. doi: 10.1200/JCO.2007.14.5466. Epub 2009 Feb 2. PMID 19188680
- [Background] Zhou C, Wu YL, Chen G, Liu X, Zhu Y, Lu S, Feng J, He J, Han B, Wang J, Jiang G, Hu C, Zhang H, Cheng G, Song X, Lu Y, Pan H, Zheng W, Yin AY. BEYOND: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Study of First-Line Carboplatin/Paclitaxel Plus Bevacizumab or Placebo in Chinese Patients With Advanced or Recurrent Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Jul 1;33(19):2197-204. doi: 10.1200/JCO.2014.59.4424. Epub 2015 May 26. PMID 26014294
- [Background] Nadler E, Yu E, Ravelo A, Sing A, Forsyth M, Gruschkus S. Bevacizumab treatment to progression after chemotherapy: outcomes from a U.S. community practice network. Oncologist. 2011;16(4):486-96. doi: 10.1634/theoncologist.2010-0287. Epub 2011 Mar 25. PMID 21441299
- [Background] Wozniak AJ, Moon J, Thomas CR Jr, Kelly K, Mack PC, Gaspar LE, Raben D, Fitzgerald TJ, Pandya KJ, Gandara DR. A Pilot Trial of Cisplatin/Etoposide/Radiotherapy Followed by Consolidation Docetaxel and the Combination of Bevacizumab (NSC-704865) in Patients With Inoperable Locally Advanced Stage III Non-Small-Cell Lung Cancer: SWOG S0533. Clin Lung Cancer. 2015 Sep;16(5):340-7. doi: 10.1016/j.cllc.2014.12.014. Epub 2015 Jan 9. PMID 25703100
- [Background] Spigel DR, Hainsworth JD, Yardley DA, Raefsky E, Patton J, Peacock N, Farley C, Burris HA 3rd, Greco FA. Tracheoesophageal fistula formation in patients with lung cancer treated with chemoradiation and bevacizumab. J Clin Oncol. 2010 Jan 1;28(1):43-8. doi: 10.1200/JCO.2009.24.7353. Epub 2009 Nov 9. PMID 19901100